CLINICAL TRIAL: NCT06632028
Title: THE EFFECT OF ARTIFICIAL INTELLIGENCE ASSISTED SPINE REHABILITATION ON GENERAL HEALTH, ANXIETY AND DISABILITY IN PATIENTS WITH CERVICAL DISC HERNIA
Brief Title: Artificial Intelligence Assisted Spine Rehabilitation in Cervical Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, SENA NUR KESKİN, physiotherapist, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OU-FTR-SNK-01
Record Dates: First submitted 2024-10-07; First posted 2024-10-08 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Herniated Intervertebral Disc
Keywords: cervical disc herniation; artificial intelligence assisted spinal rehabilitation; traditional physiotherapy; pain; general health; Anxiety; disability; herniated intervertebral disc
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: In total, two different groups will be treated. One group will receive spinal rehabilitation supported by artificial intelligence, while the other group will receive traditional physiotherapy applications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stimawell (Active Comparator): In the treatment programme to be applied to the spinal rehabilitation group supported by artificial intelligence, the patient's treatment card is first created. Artificial intelligence assisted spinal rehabilitation group will be applied 3 times a week, a total of 6 sessions and 30 minutes of treatment. The person is first prepared by lying on his back on the stimulation mat. There are 12 channels and 24 electrodes in artificial intelligence assisted spinal rehabilitation. The stimulation wave travels in all 12 L-sized channels of the stimulation mat. The two sub-channels in the M dimension are not active, the wave travels over only 10 channels. In size S only 8 channels are used, therefore 4 sub-channels of the stimulation mat are not active Artificial intelligence-assisted spinal rehabilitation overcomes skin resistance more easily with mid-frequency currents in the 2000 - 6000 Hz range compared to currents in lower frequency ranges.
  Interventions: Other: artificial intelligence assisted spinal rehabilitation; Other: conventional therapy
- convention (Other): In the traditional treatment group, a total of 15 sessions, 5 times a week, and in each session, 20 minutes of TENS application with the conventional method by placing electrodes on the painful points of the person, 20 minutes of hotpack application and 4 minutes each on the right and left sides of the neck area with intermittent ultrasound 1.5 MHz wave will be applied for a total of 8 minutes. Cervical isometric exercises will be given and 2 sets of 10 repetitions will be performed with 5 sec stretching.
  Interventions: Other: artificial intelligence assisted spinal rehabilitation; Other: conventional therapy

INTERVENTIONS:
Other: artificial intelligence assisted spinal rehabilitation — In artificial intelligence-based rehabilitation, it is more advantageous compared to other treatment methods in terms of the fact that technology applications can be designed according to the level and abilities of the individual and that the parameters such as duration, intensity, difficulty and speed of the treatment can be flexibly configured for the therapist and the patient.
Other: conventional therapy — In cervical disc herniation, non-invasive physical therapy applications such as laser treatment, hot-cold treatment methods, Transcutaneous Electrical Nerve Stimulation (TENS), interferential currents, manual therapy applications, kinesiological taping and exercise therapy, as well as painkillers and nonsteroidal anti-inflammatory drugs and antidepressive drugs are among the most preferred methods in treatment.(6)

SUMMARY:
The aim of this study is to investigate the effect of artificial intelligence-assisted spinal rehabilitation in neck hernia compared to traditional methods.

DETAILED DESCRIPTION:
Cervical disc herniation is the displacement of the intervertebral disc or nucleus pulposus in the direction of the cervical spinal canal and the resulting clinical picture. Cervical disc herniation occurs especially after the age of 40 years with disc degeneration and deterioration of the natural structure of bones and joints . Symptoms vary depending on the affected level, size and localisation of the herniation (central, lateral or foraminal). Radiculopathy accompanied by neck pain, pain radiating to the arm, paresthesia and sensory, motor and reflex changes are frequently observed . Neck pain and stiffness may radiate to the shoulder and arm. The most common complaint is neck pain, followed by paresthesia, radicular pain and weakness. It has been reported that pain originating from C6-C7 is felt in the lower part of the scapula, while pain originating from C5-C6 is felt in the middle of the medial scapula. Pain originating from C4-C5 is felt around the spine and superior to the scapula, and pain originating from C3-C4 is felt at the spinous process of the C7 vertebra and the posterior edge of the trapezius muscle. In physical examination of individuals with cervical pain due to cervical disc herniation, differences were found in ROM values, muscle strength test results, postural evaluation data, quality of life and depression levels and functional level of the neck compared to normal individuals. In cervical disc herniation, non-invasive physical therapy applications such as laser treatment, hot-cold treatment methods, Transcutaneous Electrical Nerve Stimulation (TENS), interferential currents, manual therapy applications, kinesiological taping and exercise therapy as well as painkillers and nonsteroidal anti-inflammatory drugs and antidepressive drugs are the most preferred methods in treatment. Cervical disc herniation may cause pain and various neurological deficits due to biochemical, vascular and anatomical changes in the intervertebral disc, which are influenced by extrinsic, intrinsic and genetic factors, and which occur especially as a result of exposure of the cervical region to mechanical stress. Neck pain can often be accompanied by many problems such as stiffness in the neck, headache, unilateral or bilateral shoulder pain, ocular and vestibular dysfunction.Pain caused by cervical disc herniation negatively affects the quality of life of the person.The decrease in mobility in the person with pain negatively affects physical performance, causing the person to experience inadequacies in daily life activities and decreased quality of life. In such patients, long-term imbalances between sympathetic and parasympathetic lead to various symptoms in the body. The advantages of technology applications in artificial intelligence-based rehabilitation are that it can be designed in accordance with the level and abilities of the individual, providing flexible configuration of parameters such as duration, intensity, difficulty and speed of the treatment for the therapist and patient, providing objective data with reliable and valid user detection equipment, providing real-time feedback, providing ease of activity training with real-life simulation, and reducing the possible burnout of the patient and therapist during the rehabilitation process. Conservative physiotherapy methods applied in physiotherapy have not been able to reduce the pain and participation in daily life. With artificial intelligence-assisted spinal rehabilitation, it is aimed to reduce pain and muscle spasm by determining the body calibration of individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 40-65 years old
2. Volunteering to participate in the study
3. No history of operated cervical disc herniation
4. Pain of 4 or more according to the numeric pain scale in the last 6 months

Exclusion Criteria:

1. Trauma or operation in the cervical region
2. Doing regular exercise
3. Regular use of psychiatric medication
4. Having known neurological, autoimmune diseases
5. Those who have a wound or infection in the area to be treated
6. Those with a pacemaker

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-10-04 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Informed consent form (Appendix 1), sociodemographic assessment form (Appendix 2), Numeric Pain Scale for pain severity (Appendix 3), Notham Health Profile Questionnaire for general health assessment (Appendix 4), Beck Anxiety Index for anxiety (Appendix | Conventional physiotherapy group will last for 3 weeks with 15 sessions 5 days a week, treatment duration is 1 hour. Artificial intelligence supported spinal rehabilitation will be arranged for 6 sessions 3 days a week for half an hour. Evaluations will
  In the 11-question form prepared in line with the literature, information such as personal information, contact information, medications used and whether the patient has undergone any operation are questioned. Numeric Pain Scale (NAS), which is one of the methods commonly used to determine the severity of pain, is a valid and reliable scale used to measure all pain intensities. The Beck Anxiety Scale consists of 21 questions and is used to indicate the anxiety level of individuals aged 12 years and over. Copenhagen Neck Functionality Disability Scale is a 15-item scale that measures the severity of pain and the effect of pain severity on disability in daily activities, social interaction and recreational activities and measures the person's perception of the effect of neck pain on the future. Nottingham Health Profile NSP is a general quality of life questionnaire that measures the person's perceived health problems and the extent to which these problems affect normal daily activitie

CONTACTS AND LOCATIONS:
Locations (1):
- Iskenderun Gelişim Hastanesi, Hatay, iskenderun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
When the study is finalised, researchers who want to use my data can send me an e-mail and use my data.

REFERENCES:
- [Background] Johnson JP, Masciopinto JE. Cervical-disk herniation. N Engl J Med. 1998 Sep 17;339(12):852; author reply 853. No abstract available. PMID 9750087
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9750087/